CLINICAL TRIAL: NCT04926142
Title: Prevalence of Atrial Fibrillation in Cryptogenic Stroke With Patent Foramen Ovale Closure (PFO-AF) Study
Acronym: PFO-AF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A03417-32
Record Dates: First submitted 2021-06-11; First posted 2021-06-14 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Patent Foramen Ovale; Atrial Fibrillation; Stroke
MeSH Terms: conditions — Foramen Ovale, Patent; Atrial Fibrillation; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients planned for percutaneous PFO closure: Patients will undergo implantation of a Holter device (Reveal Linq Medtronic) 2 months prior to percutaneous PFO closure. Devices will be monitored by telemonitoring until the PFO closure procedure, and at 2, 12 and 24 months after the procedure.
  Interventions: Device: Implantation of Holter device; Procedure: Percutaneous PFO closure

INTERVENTIONS:
Device: Implantation of Holter device — Implantation of a Holter device (Reveal Linq, Medtronic) for telemonitoring of cardiac rhythm
Procedure: Percutaneous PFO closure — Patients will undergo percutaneous closure of patent foramen ovale

SUMMARY:
This study aims to assess the incidence of atrial fibrillation (AF), documented using data recorded by an implantable Holter monitoring device (Reveal Linq, Medtronic) within 2 years after percutaneous closure of patent foramen ovale for cryptogenic stroke.

DETAILED DESCRIPTION:
This study aims to assess the incidence of atrial fibrillation (AF), documented using data recorded by an implantable Holter monitoring device (Reveal Linq, Medtronic) within 2 years after percutaneous closure of patent foramen ovale (PFO) for cryptogenic stroke. Secondary objectives include assessment of the burden of AF at 2, 12 and 24 months after PFO closure; evaluation of the relationship between plasma levels of MR proANP and presence of AF within 2 years after percutaneous PFO closure in patients with a history of cryptogenic ischemic stroke; and description of recurrence rates for stroke (ischemic and hemorrhagic), major bleeding, minor bleeding, peripheral emboli during the 2-year follow-up period after percutaneous PFO closure, in patients with and without AF.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged >18 years)
* with an indication for percutaneous closure of PFO due to cryptogenic stroke, with indication validated by a cardio-neurological team.
* patients must provide written informed consent
* patients must be affiliated to a social security regime or be a beneficiary thereof.

Exclusion Criteria:

* Patients under legal protection
* Patients not affiliated to any social security regime
* Patients within the exclusion period of another clinical trial as per the national registry of research volunteers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective patients who have had cryptogenic stroke (ischemic only) and with patent foramen ovale confirmed by transoesophageal echocardiography, with an indication for percutaneous closure.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2025-08-21 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation | Within 2 months after percutaneous PFO closure
  Occurrence of documented atrial fibrillation (i.e. at least one episode lasting 30 seconds)

SECONDARY OUTCOMES:
Atrial fibrillation | Within 24 months after percutaneous PFO closure
  Occurrence of documented atrial fibrillation (i.e. at least one episode lasting 30 seconds)
Burden of atrial fibrillation | Within 2 years after percutaneous PFO closure
  Cumulative total time in atrial fibrillation (in days, hours, minutes)
Relation between MR proANP levels and atrial fibrillation | Within 2 years after percutaneous PFO closure
  Relation between pre-procedure circulating venous MR proANP levels and atrial fibrillation defined as per the primary endpoint
Stroke | Within 2 years after percutaneous PFO closure
  Ischemic or hemorrhagic stroke documented by CT or MRI
Peripheral emboli | Within 2 years after percutaneous PFO closure
  Peripheral emboli by CT or MRI
Bleeding | Within 2 years after percutaneous PFO closure
  Major or minor bleeding according to the ISTH classification

CONTACTS AND LOCATIONS:
Overall Officials: Marc Badoz, MD, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (4):
- France (4):
  - University Hospital Besancon, Besançon
  - CHU Lyon - Hôpital Louis Pradel, Bron
  - CHU Dijon, Dijon
  - CHU Grenoble, Grenoble

REFERENCES:
- [Derived] Badoz M, Derimay F, Serzian G, Besutti M, Rioufol G, Frey P, Guenancia C, Ecarnot F, Meneveau N, Chopard R. Incidence of atrial fibrillation in cryptogenic stroke with patent foramen ovale closure: protocol for the prospective, observational PFO-AF study. BMJ Open. 2023 Sep 12;13(9):e074584. doi: 10.1136/bmjopen-2023-074584. PMID 37699623